CLINICAL TRIAL: NCT06839898
Title: A Prospective, Randomized Clinical Study of Two Phakic Toric Implantable Lenses to Compare Outcomes in Patients With Moderate to High Myopia and Astigmatism
Brief Title: A Prospective, Randomized Clinical Study of Two Phakic Toric Implantable Lenses
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biotech Healthcare Holding Gmbh (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BTVCPL-PHAKICTORIC-2019-13; CIV- 20-09-034764 (Other: EUDAMED)
Record Dates: First submitted 2025-01-09; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Myopia, Moderate; Myopic Astigmatism; Myopia, Degenerative
MeSH Terms: conditions — Myopia; Lymphoma, Follicular; Astigmatism; Myopia, Degenerative

STUDY DESIGN:
Intervention Model Description: Phakic intraocular lenses are clear implantable lenses that are surgically placed either in anterior chamber (AC) or posterior chamber (PC) without removing the natural lens, enabling light to focus on the retina for improved uncorrected visual acuity. Phakic intraocular lenses demonstrate high optical quality and potential gain in visual acuity in myopic patients due to retinal magnification. Toric version of phakic intraocular lens is intended to correct both myopia and astigmatism
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EYECRYLTM Phakic Toric Intraocular Lens Treatment Arm (Experimental): Patients will be implanted with Eyecryl Phakic Toric IOL based on randomization.
  Interventions: Device: EYECRYLTM Phakic Toric Intraocular Lens Treatment Arm
- Visian® Toric ICL Treatment Arm (Active Comparator): Patients will be implanted with Visian® Toric ICL based on randomization.
  Interventions: Device: Visian® Toric ICL Treatment Arm

INTERVENTIONS:
Device: EYECRYLTM Phakic Toric Intraocular Lens Treatment Arm — The patients will be implanted with Eyecryl Phakic IOL at this arm based on randomization.Phakic intraocular lenses are clear implantable lenses that are surgically placed either in anterior chamber (AC) or posterior chamber (PC) without removing the natural lens, enabling light to focus on the retina for improved uncorrected visual acuity. Phakic intraocular lenses demonstrate high optical quality and potential gain in visual acuity in myopic patients due to retinal magnification. Toric version of phakic intraocular lens is intended to correct both myopia and astigmatism.
  Arms: EYECRYLTM Phakic Toric Intraocular Lens Treatment Arm
Device: Visian® Toric ICL Treatment Arm — The patients will be implanted with Visian® Toric Implantable Contact Lens at this arm based on randomization. Phakic intraocular lenses are clear implantable lenses that are surgically placed either in anterior chamber (AC) or posterior chamber (PC) without removing the natural lens, enabling light to focus on the retina for improved uncorrected visual acuity. Phakic intraocular lenses demonstrate high optical quality and potential gain in visual acuity in myopic patients due to retinal magnification. Toric version of phakic intraocular lens is intended to correct both myopia and astigmatism.
  Arms: Visian® Toric ICL Treatment Arm

SUMMARY:
Primary Objective: To compare the efficacy and the residual refractive error of EYECRYLTM Phakic toric versus Visian® Toric ICL in moderate to high myopic patient with co-existing astigmatism. Secondary Objectives: To evaluate and compare the safety of EYECRYLTM Phakic toric versus Visian® Toric ICL in moderate to high myopic patients with co-existing astigmatism.

DETAILED DESCRIPTION:
Phakic intraocular lenses are clear implantable lenses that are surgically placed either in anterior chamber (AC) or posterior chamber (PC) without removing the natural lens, enabling light to focus on the retina for improved uncorrected visual acuity. Phakic intraocular lenses demonstrate high optical quality and potential gain in visual acuity in myopic patients due to retinal magnification. Toric version of phakic intraocular lens is intended to correct both myopia and astigmatism.1

ELIGIBILITY:
Inclusion Criteria:

* Patients 21 years old or older.
* Calculated IOL Power is within the range of the investigational IOLs
* Corneal Cylindrical error within the range defined in the clinical investigation plan
* Subject has monocular UCVA 0.5 LogMAR or worse
* Subject has had a stable refraction (±0.5D; ±1.0D for higher refractive errors), as expressed by manifest refraction spherical equivalent (MRSE) for a minimum 12 months prior to surgery, verified by consecutive refractions and/or medical records or prescription history.
* Subject, who is a current contact lens wearer, needs to demonstrate a stable refraction (±0.5D) expressed as MRSE, on two consecutive examination dates and stability of the refraction is determined by the following criteria:

  1. Contact lenses were not worn for at least 2 weeks or 3 days prior to the first refraction.
  2. Two refractions were performed at least 7 days apart.
* Subject, who is expected to have residual postoperative cylindrical refractive error of ≥1D, has been given the opportunity to experience his/her best spectacle vision with the anticipated correction.
* Expected dilated pupil size at least large enough to visualize the axis marking.
* Patients willing to attend all follow-up appointments
* Patients must sign and be given a copy of the written Informed Consent form

Exclusion Criteria:

* Subject with acute and chronic disease or illness that would increase the operative risk or confound the outcomes of the evaluation.
* Subject taking systematic medication that can confound the outcome of the study or increase the risk to the subject
* Subject with ocular condition that may predispose the subject to future complications
* Subject with previous intraocular or corneal surgery
* Subject with less than the minimum endothelial cell density 2000 cells/mm² at the time of enrollment
* Pregnant or planning to become pregnant, or is lactating during the course of the evaluation
* Other condition associated with fluctuation of hormones
* ACD measured from the endothelium lower than 2.8 mm
* Concurrent participation in another drug or device evaluation.
* Any cataract of any grade.
* Coefficient of variation of endothelial cell area >0.45
* Percent Hexagonality of endothelial cell shape ≤ 45%
* Monocular subject
* Vulnerable subjects as defined in section 12.3.10

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2021-10-10 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
The mean residual refractive error | 6 Month
  The mean residual refractive error in the study lens population that is equivalent to the mean residual refractive error of the control lens within +/- 0.50 Diopters at the 6-months post-op visit.

CONTACTS AND LOCATIONS:
Locations (4):
- Germany (3):
  - Precise Vision Augentagesklinik Greven, Münster, North Rhine-Westphalia
  - Precise Vision Augentagesklinik Rheine, Rheine, North Rhine-Westphalia
  - Precise Vision Augentagesklinik Rheine, Steinfurt, North Rhine-Westphalia
- Netradhama Superspeciality Eye Hospital, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: No